CLINICAL TRIAL: NCT04482985
Title: Meclizine Plasma Levels in Responders and Non-responders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Yoni Gutkovich, deputy of the head of department for the human performance laboratory, the Israeli naval institute, Haifa., Medical Corps, Israel Defense Force
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2019
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Seasickness; Meclizine
Keywords: Seasickness; Plasma Levels; Meclizine
MeSH Terms: conditions — Motion Sickness | interventions — Meclizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Meclizine responders (Active Comparator)
  Interventions: Drug: Meclizine Hydrochloride
- Meclizine non responders (Active Comparator)
  Interventions: Drug: Meclizine Hydrochloride

INTERVENTIONS:
Drug: Meclizine Hydrochloride — Meclzine is given to all study participants to prevent seasickness. Meclizine plasma levels are determined from both the meclizine responders and non responders group.
  Other Names: Bonine

SUMMARY:
Motion sickness is a debilitating condition that can effect many crew members. Meclizine has long been known as an effective anti motion sickness drug. The response to the drug is variable - some are responders, while others are resistant to the drug. The aim of the present study is to examine whether there is a correlation between meclizine plasma levels and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Seasickness questioner (WIKER) score of 7.
* Subjective functioning at 1 meter sea voyage - 5/10 and lower.
* Subjects who were prescribed 25mg of meclizine.
* Subjects who did not take any other drugs 48 prior to their participation in the study.

Exclusion Criteria:

* Known hearing loss or any vestibular impairment
* Vertigo complains
* Any ear infection
* Use of Scopolamine based anti-seasickness drugs.
* Use of meclizine 50mg.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Meclizine plasma levels | 2 hours after meclizine administration
  ng/dl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Qian S, Zhang Q, Chow MS. Quantification of meclizine in human plasma by high performance liquid chromatography-mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Jan 1;879(1):95-9. doi: 10.1016/j.jchromb.2010.11.022. Epub 2010 Dec 1. PMID 21163711